CLINICAL TRIAL: NCT06954506
Title: The Effect of Reiki on Hopelessness Level in Oncology Patients Receiving Chemotherapy Treatment; Randomised Controlled Trial
Brief Title: The Effect of Reiki on Hopelessness Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Reiki and Oncology Patients; Reiki and Oncology Patients (Registry Identifier: Reiki and Oncology Patients)
Record Dates: First submitted 2025-04-07; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Oncology Patients
Keywords: Reiki; oncology; hopelessness
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The research data were collected using the "Individual Information Form" and the "Beck Hopelessness Scale" through face-to-face and telephone interviews after obtaining ethical committee approval. The time required for individuals to complete the forms is approximately 10 minutes. Patients were informed about the application, and a Reiki application video prepared/selected by the researchers was shared with the patients. Patients were asked to perform Reiki every day for a week following each chemotherapy session for 4 cycles. A reminder message was sent to the patients the day before each cycle for the Reiki application. The level of hopelessness was reassessed at the end of each week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki Group (Experimental): Patients were informed about the application, and a Reiki application video prepared/selected by the researchers was shared with the patients. Patients were asked to perform Reiki every day for a week following each chemotherapy session for 4 cycles. A reminder message was sent to the patients the day before each cycle for the Reiki application. The level of hopelessness was reassessed at the end of each week.
  Interventions: Behavioral: Reiki Group
- control group (No Intervention): Only data collection forms were filled in the control group. No intervention was made.

INTERVENTIONS:
Behavioral: Reiki Group — Patients were informed about the application, and a Reiki application video prepared/selected by the researchers was shared with the patients. Patients were asked to perform Reiki every day for a week following each chemotherapy session for 4 cycles. A reminder message was sent to the patients the day before each cycle for the Reiki application. The level of hopelessness was reassessed at the end of each week.
  Arms: Reiki Group

SUMMARY:
This quasi-experimental study aims to examine the effect of Reiki on the level of hopelessness in oncology patients.

The study was conducted at İzmir Tepecik Training and Research Hospital with 32 patients in both experimental and control groups. Patients performed Reiki daily for a week following each chemotherapy session for 4 cycles. Data were collected using the "Individual Information Form" and the "Beck Hopelessness Scale" through face-to-face and telephone interviews. Ethical approval was obtained, and data were analyzed using SPSS.

DETAILED DESCRIPTION:
Reiki is considered a complementary and alternative therapy method that can be effective in coping with such emotional challenges and enhancing psychological well-being. It is thought that Reiki practices, by regulating the flow of energy and providing deep relaxation, can reduce individuals' levels of hopelessness and improve overall quality of life. This study will investigate the effect of Reiki practices on the levels of hopelessness in oncology patients.

ELIGIBILITY:
inclusion criteria: Receiving treatment at the Outpatient Chemotherapy Unit of İzmir Tepecik Training and Research Hospital University of Health Sciences, Diagnosed with cancer, Aged 18 and over, Willing to participate in the research

exclusion criteria: Not willing to participate in the research, Having communication problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
The research data will be collected using the "Individual Information Form" and the "Beck Hopelessness Scale" prepared by the researchers in line with the literature. | The research data were collected through face-to-face and telephone interviews after obtaining ethical committee approval. The time required for individuals to complete the forms is approximately 10 minutes.
  Individual Information Form: The form prepared by the researchers consists of 14 questions.
  Beck Hopelessness Scale: The Beck Hopelessness Scale was developed by Beck and colleagues in 1974 to determine the degree of pessimism an individual has about the future. The scale consists of 20 items in a five-point Likert format. The questions are answered as true or false and reflect negative expectations. Each answer that matches the given key scores 1 point, while answers that do not match score 0 points. The total score obtained is considered the "hopelessness" score, with higher scores indicating higher levels of hopelessness. The scale's score range is 0-20. The questions on the scale cover emotional, motivational, and cognitive dimensions. The scale consists of three factors: "Feelings about the Future," "Loss of Motivation," and "Future Expectations" (Durak & Palabıyıkoğlu, 1994). In this study, the Cronbach's Alpha value for hopelessness was calculated as 0.952.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze TEMİZ, Dr, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Health Science University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No